CLINICAL TRIAL: NCT00122733
Title: Facilitation of Weaning From Ventilator by Loxapine
Brief Title: Loxapine and Weaning From Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMR2
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Respiratory Insufficiency; Psychomotor Agitation
Keywords: Mechanical ventilation; Agitation; Difficult weaning
MeSH Terms: conditions — Respiratory Insufficiency; Psychomotor Agitation | interventions — Loxapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: loxapine

SUMMARY:
Patients may be very agitated during the weaning period from mechanical ventilation. Administration of loxapine, a neuroleptic that does not notably affect ventilatory drive, may help in obtaining an adequate level of cooperation and, therefore, in reducing the duration of mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation is a life-saving procedure in critically ill patients. This procedure is however not devoid of risks and every effort should be made to shorten its duration. This is best accomplished by the implementation of weaning protocols. Sedation (by opiates and benzodiazepines) is often required in such patients for their comfort and adaptation to the respirator. Withdrawal of sedation in order to allow patients to resume spontaneous breathing may be associated with agitation and confusion that may hinder weaning. In such cases, reinstitution of heavy sedation will prolong ventilator-dependency. It may therefore be interesting to administer a neuroleptic (loxapine) with good anxiolytic properties but that does not notably interfere with spontaneous breathing ability.

Patients will be included when they fail a spontaneous ventilation trial (see inclusion criteria) because of marked agitation. Usual simple clinical (respiratory frequency, P01 measured on the respirator, arterial pressure, cardiac rate) and biological criteria (arterial blood gas determination) and a measurement of sedation/agitation with validated scales (Richmond agitation sedation scale, Ramsay score) will be gathered when a patient is deemed ready for a trial of spontaneous ventilation for weaning. In cases of marked agitation according to validated scales, patients will be given a conventional dose (150 mg) of loxapine by the nasogastric tube and the efficacy of this treatment will be evaluated on the same parameters as above. Demonstration of the facilitation of weaning by this simple strategy would be useful in order to reduce risks associated with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for weaning from the respirator (FIO2 less than 50%; positive end expiratory pressure [PEEP] level less than 6 cmH2O)
* Patients whose agitation (according to accepted scores) during a weaning trial precludes extubation

Exclusion Criteria:

* History of convulsions or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
cessation of agitation | 3 hours
improvement in the clinical and biological parameters of weaning trial | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHEVREL, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Réanimation, Hopital Louis Mourier, Colombes, France

REFERENCES:
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Truman B, Ely EW. Monitoring delirium in critically ill patients. Using the confusion assessment method for the intensive care unit. Crit Care Nurse. 2003 Apr;23(2):25-36; quiz 37-8. No abstract available. PMID 12725193